CLINICAL TRIAL: NCT01210066
Title: Pain, Opioids and Pro-Inflammatory Immune Responses
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit prescription opioid abusers; ultimately no potential POA recruit passed the pre-screening process
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 5R21DA027558 (NIH)
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Pro-inflammatory Activity; Immunologic Activity Alteration
Keywords: inflammation; opioid-induced hyperalgesia; bupenorphine; prescription opioid abuse
MeSH Terms: conditions — Inflammation; Opioid-Related Disorders | interventions — Fentanyl; Analgesics, Opioid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pain Challenge (Active Comparator): Cold pressor test
  Interventions: Other: Cold pressor test
- Pain + Opioid Challenge (Active Comparator): IV fentanyl 1mcg/kg followed by cold pressor test
  Interventions: Other: Fentanyl plus cold pressor test
- Opioid Challenge (Active Comparator): Administration of fentanyl 1mcg/kg of subject weight
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — IV fentanyl 1mcg/kg
  Other Names: opioid
  Arms: Opioid Challenge
Other: Cold pressor test — Non-dominant arm submerged in ice water (0 degrees Celsius) until it is no longer tolerable but less than 5 minutes
  Other Names: cold pressor task
  Arms: Pain Challenge
Other: Fentanyl plus cold pressor test — fentanyl IV 1mcg/kg fifteen minutes prior to cold pressor test (arm submerged in ice water until no longer tolerable but no longer than 5 minutes)
  Other Names: opioid and cold pressor
  Arms: Pain + Opioid Challenge

SUMMARY:
Providing pain management to the patient who abuses prescription opioids presents a clinical challenge, not only due to concerns about "drug-seeking", but because they have increased sensitivity to pain, a phenomenon identified as opioid-induced hyperalgesia (OIH). In an effort to improve pain treatment, the aims of the proposed work are to evaluate the analgesic and hyperalgesic effects of opioids to acute pain in this vulnerable population, and to examine the role of opioid-induced proinflammatory changes in these responses.

DETAILED DESCRIPTION:
Both acute pain and opioid administration have been shown to induce a systemic pro-inflammatory response. However, the presence of these inflammatory responses is unknown in situations where a co-occurrence of pain and opioid administration exists as is the common clinical case of a patient with acute pain and taking opioid analgesics. A patient population for whom the combined effects of pain and opioids on immune function are particularly complex are the estimated 5.2 million Americans aged 12 or older who abuse prescription opioids. Not only are these individuals at risk for poor pain management due to their status as an "addict", but there is good preclinical evidence to suggest that their chronic opioid use brings with it a general state of systemic inflammation, and thus setting the patient up for a unique or enhanced inflammatory response to the combination of acute opioids and pain. To better understand the health implications of treating acute pain with opioids in patients and in particular, those who abuse prescription opioids, inflammatory responses to the main and interaction effects of acute pain and opioid administration will be examined in well-characterized samples of each. Specifically, we will evaluate the inflammatory and cytokine responses to: (1) experimental pain; (2) an acute opioid challenge; and (3) the combination of opioid administration followed by cold-pressor pain, in healthy control subjects and age- and gender-matched prescription opioid abusers.

ELIGIBILITY:
Inclusion criteria:

* male and non-pregnant female, non-smoking adults in good general health
* between the ages of 21-40 years old
* fluent in English with willingness to participate in the research study

Supplementary Inclusion Criteria: Prescription Opioid Abusers

* DSM-IVR diagnosis of prescription opioid abuse or dependence disorder
* compliance in treatment and on a stable dose of buprenorphine (6-24mg/day) x at least 10 days prior to screening
* Participation in an ISAP treatment program or a qualified community-based opioid treatment program or private clinic for the entire duration of their study participation

Exclusion criteria:

* regular use of any medication that influences immune status or immune system function
* regular use of a medication that influences pain perception, including opioids (* only for healthy subjects population*)
* Regular use of a medication that influences pain perception, except for buprenorphine (** only for POA population**)
* known hypersensitivity to opioids or no previous opioid exposure (*only healthy controls)
* presence of acute or chronic pain syndrome
* neuropsychiatric illness (i.e., peripheral neuropathy, schizophrenia) known to affect pain perception
* presence of chronic immune compromise (hepatitis C, HIV) or acute infection within the last four weeks
* current or past history of high blood pressure, heart disease, or stroke, or currently have a pacemaker.
* current DSM-IV diagnosis
* BMI less than 18.5 or greater than 29.9
* History of sleep apnea

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
plasma levels of pro-inflammatory cytokine IL-6 | 15 minutes prior to fentanyl administration, 60 and 180 minutes post fentanyl administration,
  inflammatory cytokine activity will be evaluated with an in vivo approach over a three hour period of time to enable observation of the duration of opioid activity

CONTACTS AND LOCATIONS:
Overall Officials: Peggy A Compton, RN PhD FAAN, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA School of Nursing, Los Angeles, California, United States

REFERENCES:
- [Result] Compton P, Griffis C, Breen EC, Torrington M, Sadakane R, Tefera E, Irwin MR. Opioid treatment of experimental pain activates nuclear factor-kappaB. J Opioid Manag. 2015 Mar-Apr;11(2):115-25. doi: 10.5055/jom.2015.0261. PMID 25901477